CLINICAL TRIAL: NCT06933186
Title: NEUROPSYCHOLOGICAL REHABILITATION OF EXECUTIVE FUNCTIONS IN ALCOHOL USE DISORDER: RANDOMIZED PILOT CLINICAL TRIAL PROTOCOL
Brief Title: NEUROPSYCHOLOGICAL REHABILITATION FOR ALCOHOL USE DISORDERS
Acronym: AUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: ULSSJOSÉ (Unknown)
Responsible Party: Principal Investigator, Sónia Ferreira, Psychologist- Principal Investigator, University of Lisbon
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105/21
Record Dates: First submitted 2025-03-13; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder Cognitive Decline
Keywords: Executive functioning; Neuropsychological Rehabilitation; Alcohol Use Disorder; Working memory; Inhibition; Cognitive Flexibility; Planning
MeSH Terms: conditions — Alcoholism; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Two-arm pilot clinical trial; two groups (control and experimental), with different interventions, compared at the same time, to evaluate the effectiveness of neuropsychological rehabilitation
Who Masked: Investigator
Masking Description: To ensure that the attribution of interventions is hidden from researchers, the collaboration of a nursing member, not involved in the research, will be used to carry out the random distribution of the sample, using a random number generator, after recruitment and the first assessment. A psychologist will be included to exclusively carry out the Neuropsychological Rehabilitation program. The collection, recording, processing and analysis of data from the different phases of the research collection process will be exclusive to the researcher, and the anonymization of participants and the non-identification of group allocation will be guaranteed until the end of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Other): This group, in addition to weekly therapeutic groups (usual treatment), will attend neuropsychological rehabilitation. This will last for 3 months, starting after alcohol detoxification, three times a week. It includes three components: cognitive training, psychoeducation and social skills/emotional management training. The cognitive training consists of 36 sessions, each lasting approximately 1h30 and will focus on the various components of EF (basic EF: working memory, inhibition, cognitive flexibility and complex functions: planning) and other cognitive domains (attention, memory, language), including different pencil and paper exercises and an online cognitive training platform Cogweb (Neuroinova, 2007), in which the exercises progress automatically through levels, becoming progressively more difficult.
  Interventions: Behavioral: Neuropsychological rehabilitation; Behavioral: Weekly therapeutic groups
- Control Group (Other): The control group will attend weekly therapeutic groups, which consist of open groups, aimed to promote abstinence and relapse prevention, supporting the management of difficulties in the person's daily life related to consumption, promoting psychoeducation about the disease and coping strategies to deal with craving. At the end of the investigation, the possibility of completing the RN program will be made available to all participants in the control group, which the experimental group accessed.
  Interventions: Behavioral: Weekly therapeutic groups

INTERVENTIONS:
Behavioral: Neuropsychological rehabilitation — Neuropsychological rehabilitation includes an integrated approach, consisting of three components: cognitive training; psychoeducation; and social skills/emotional management training. Cognitive training uses a combination of different tasks (always covering attention, memory and executive functions exercises), with a 30-minute session on the online cognitive training platform and 1 hour of pencil and paper exercises in a group, in a total of 36 sessions . Psychoeducation addresses specific topics related to Alcohol Use Disorder and its cognitive impact. Social skills/emotional management training includes problem-solving exercises, assertiveness training, emotion identification and management, among others. These sessions will be held once a week, for a total of 12 sessions.
  Arms: Experimental Group
Behavioral: Weekly therapeutic groups — The control group will attend weekly therapeutic groups, which consist of open groups, aimed to promote abstinence and relapse prevention, supporting the management of difficulties in the person's daily life related to consumption, promoting psychoeducation about the disease and coping strategies to deal with craving

SUMMARY:
This investigation will take place between September 2024 and June 2025, with the objective of analyzing executive deficits and the impact of Neuropsychological Rehabilitation on Alcohol Use Disorder, comparing different evaluation moments. Data will be collected at UTRA and Clinica 4, at ULSSJOSÉ, from a total of 48 participants at the end of three months, using a semi-structured interview, in order to obtain sociodemographic data and information related to alcohol consumption, as well as the application of a set of clinical and neuropsychological tests. This first assessment will be carried out after medically assisted detoxification (from the 10th day of abstinence), and subsequently the participants will be randomly distributed into two groups, a control group that will carry out the therapeutic groups (usual treatment) and a group experimental group that, in addition to these groups, will attend the Neuropsychological Rehabilitation Program. All participants will be assessed again, one, three and six months after the first assessment. This research will have the benefit of structuring interventions that are more tailored to the needs of people with AUD, seeking to minimize the impact of cognitive deficits on their physical and mental health. Participation in the study will be voluntary, and the risks for participants will be non-existent. No payment will be made to participants for their collaboration in the study. The confidentiality and anonymity of participants will be guaranteed, as well as the security of personal and clinical data, safeguarding the rights and freedoms of the data holder. The data collected will be used only for this purpose, with access to them being exclusive to the researcher, who has sole responsibility for processing and publishing the data, always seeking to preserve the identity of the participants. The data will only be kept for the time necessary to carry out the purpose of the investigation.

DETAILED DESCRIPTION:
The aim is to carry out a pilot randomized clinical trial, blinded to the researchrs (from September 2024 to June 2025), with two arms: an experimental group and a control group. The experimental group will have access to the Neuropsychological Rehabilitation program and weekly therapeutic groups. The Neuropsychological Rehabilitation program will last three months and includes three components: psychoeducation, cognitive training and social skills/emotional management training. Cognitive training will use different strategies such as: pencil and paper exercises and an online cognitive training platform - Cogweb (Neuroinova, 2007). The control group will only participate in weekly therapy groups, which consist of open groups that aim to help people manage everyday difficulties related to alcohol consumption, providing psychoeducation on coping strategies to deal with cravings.Participants will be recruited from the Alcohol and New Addictions Service (inpatient) and the Alcohol Treatment and Rehabilitation Unit (outpatient), at Hospital Júlio de Matos, ULSSJOSÉ.

In the first phase, participants will be recruited in this Service, carrying out a prior analysis, taking into account the inclusion/exclusion criteria, carried out by the treatment team,and the Montreal Cognitive Assessment - MoCA (Simões, Freitas, Santana, Firmino, Martins, Nasreddine, Vilar, 2008) also being applied, to assess whether they do not present cognitive impairment. . After this recruitment, information about the study will be provided and all doubts will be clarified, to complete the informed consent. The first assessment will take place from the 10th day of abstinence. This will involve the application of a battery of tests that includes a semi-structured interview (evaluating sociodemographic information and characterization of consumption), clinical tests (evaluating degree of dependence; anxiety and depression; quality of life) and neuropsychological tests to evaluate executive functions. One month later, an assessment will be carried out, including only the Frontal Assessment Battery - FAB and a description of consumption, as a way of monitoring progress in these components. Subsequently, two evaluations will be carried out with the complete battery, described in the outcome measures, one at three months and the other at six months. Throughout the assessment sessions or intervention sessions, users will have their consumption monitored with the alcohol test.

The primary outcome was defined as performance regarding general executive functioning, assessed with the total FAB score, comparing the baseline with the result at one, three and six months, in both groups.

As secondary outcomes the investigators intend to analyze:

* Performance in working memory, cognitive flexibility, inhibition and planning, measured by scoring the letters and numbers test of the Wechsler Intelligence Scale for adults - WAIS-III, Wisconsin Card Test ,Trail Making Test- TMT, Stroop Color and Word Test, Zoo Map and Search for Keys from the Behavioral Assessment of the Dysexecutive Syndrome (BADS) , respectively, comparing the baseline with the results at three and six months, in both groups performance in other cognitive domains such as verbal fluency (verbal fluency test score) and information processing speed (code test score), measured between the two groups, after three and six months, comparing with baseline data, in both groups;
* changes in the level of alcohol consumption (analyzed through the variables number of relapses, number of detoxifications, consumption time, abstinence time in days, number of standard drinks), comparing the baseline results with those of three and six months, in both groups;
* changes in quality of life, comparing the baseline with the results at three and six months, (World Health Organization quality of life (WHOQOL) - BREF score), in both groups.
* Performance in the cognitive domains studied, comparing the results of the baseline, three and six months between genders.

In statistical terms, univariate and bivariate descriptive analysis methodologies will be applied. In the analysis of baseline results, chi-square tests will be used to study the association of qualitative variables and t-tests for independent samples or nonparametric Mann-Whitney tests to compare two groups in quantitative variables. The aim is to compare two or three evaluation moments, using t-tests for paired samples or nonparametric Friedman tests. Additionally, for each group separately, the association between the main outcome variables and the sociodemographic characteristics of the individuals will be analyzed (applying the appropriate tests for the types of variables studied). The application of mixed ANOVA with repeated measures will be considered to compare the groups across the evaluation moments. The application of Logistic Regression will also be considered using FAB performance above or equal to the threshold of 14 as a dependent variable and associating it with potential risk and protective factors (identified as relevant by bivariate analysis). A characterization of the individuals who abandon the study (dropouts) will be performed. Whenever necessary, a significance level of 5% and a confidence level of 95% will be considered.

The study was approved by the Scientific Pedagogical Committee and the Ethics Committee for Health of the institution where it will be carried out, and by the Ethics Committee of the CAML of the Faculty of Medicine of Lisbon. Results will be disseminated in peer-reviewed publications and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* People who attend the Alcoholics and New Addictions Services and the Alcoholics Treatment and Rehabilitation Unit (UTRA), of the S. José Local Unit (ULSSJosé),
* undergoing medically assisted detoxification, inpatient or outpatient.
* diagnosis of PUA; be abstinent for at least 10 days; both genders;
* sign informed consent.

Exclusion Criteria:

* no indication of cognitive deterioration in the Montreal Cognitive Assessment (MOCA ≥ 26)
* severe neurological disease (stroke; traumatic brain injury; epilepsy; alcoholic dementia; Wernicke-Korsakoff condition, major neurological condition)
* severe mental disorder (psychosis; severe personality disorder);
* consumption of other toxic substances at the time of assessment;
* age under 18;
* serious physical illness;
* acute alcohol intoxication
* refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Frontal Assessment Battery - FAB (total score) (Lima, Meireles, Fonseca, Castro, Garrett; 2008). | Baseline, one, three and six months
  * assessment general executive functioning
  * divided into six subscales: abstract thinking (test of similarities); mental flexibility (phonemic fluency); motor programming (Luria motor series - fist-edge-palm patterns); sensitivity to interference (antagonistic instructions); inhibitory control (go-no-go) and environment independence (suppression of grasping behavior);
  * minimum score: 0; maximum score: 18;
  * a higher score indicates better cognitive function;
  * cutoff point: ≥14 (without prejudice to function).

SECONDARY OUTCOMES:
Letter-number sequence subscale of the Wechsler Adult Intelligence Scale - WAIS-III (Weschler et al, 2017) | Baseline, three and six months
  * Assessment working memory
  * higher scores mean better results
  * the score is standardized considering age and level education.
Verbal Fluency Test (Cavaco et al, 2013a) | Baseline, three and six months
  * assesses the ability to generate words, considering the semantic (Semantic Verbal Fluency) and phonemic (Phonemic Verbal Fluency) categories - only the phonemic category will be used;
  * The greater the number of words produced, the better the results.
  * the data is standardized considering age and education
World Health Organization Quality of Life - BREF - WHOQOL-BREF (WHOQOL Group;1998; Skevington et al, 2004) | Baseline, one, three and six months
  * Assessment quality of life;
  * Organized into four dimensions of quality of life: physical, psychological, social relations and environment;
  * Calculation of a general quality of life indicator
  * The score ranges from 0 to 100, with a higher score corresponding to a better perception of quality of life
Trail Making Test - TMT (Cavaco et al, 2013) | Baseline, three and six months
  * Assesses cognitive flexibility;
  * Consists of two parts (A and B); only part B will be used in this investigation.
  * Time (in seconds) is counted, which the criterion is for scoring the test;
  * The longer the execution time, the worse the results
  * The data is standardized considering age and education
Stroop Color and Word Test (Fernandes, 2013) | Baseline, three and six months
  * Assessment inhibition;
  * The quote corresponds to the number of elements performed within a 45-second interval, and Interference is also calculated.
  * Normative performance corresponds to one standard deviation of the population mean.

OTHER OUTCOMES:
Severity of Alcohol Dependence Questionnaire -SADQ (Breda et al., 2018) | one, three and six months
  * Assesses the degree of alcohol dependence;
  * obtains a severity index that varies between >16 points - mild dependence; 16-30 - moderate dependence and <31 - severe dependence.
Hospital Anxiety and Depression Scale- HADS (McIntyre et al, 1999) | one, three and six months
  * Assesses emotional aspects (anxiety and depression);
  * -Minimum score: 0; maximum score: 21;
  * Higher values indicate higher levels of anxiety and depression;
  * Anxiety and depression can be classified as "normal" (0-7), mild (8-10), moderate (11-15) and severe (16-21)
Montreal Cognitive Assessment - MOCA (Simões, Freitas, Santana, Firmino, Martins, Nasreddine, Vilar; 2008) | one moth
  * Global cognitive assessment, grouped into the following dimensions: short-term memory, executive functions, visuospatial capacity, language, attention, concentration and working memory and temporal and spatial orientation;
  * Cutoff point: ≥ 26; means cognitive deterioration.
Sociodemographic questionnaire | Baseline, one, three and six months
  Sociodemographic characterization of the sample

CONTACTS AND LOCATIONS:
Overall Officials: Sónia Ferreira, MSc, Principal Investigator — Unidade de Tratamento e Reabilitação de Alcoólicos (UTRA), na Unidade de Local de São José. Lisboa; Faculdade de Medicina. Universidade de Lisboa.; Cristina Ribeiro, PhD, Study Chair — Faculdade de Medicina. Universidade de Lisboa. Lisboa; Instituto de Medicina Preventiva e Saúde Pública. Clínica Universitária de Medicina Geral e Familiar; Samuel Pombo, PhD, Study Chair — Serviço de Psiquiatria e Saúde Mental do Hospital de Santa Maria/Clinica Universitária de Psiquiatria e Psicologia Médica da Faculdade de Medicina.; Leonor Bacelar-Nicolau, PhD, Study Chair — Instituto de Saúde Ambiental e Instituto de Medicina Preventiva e Saúde Pública - Faculdade de Medicina. Universidade de Lisboa.; Enrique Vásquez-Justo, PhD, Study Chair — Escola Superior de Educação de Fafe. Braga. Universidad Camilo José Cela: Villafranca del Castillo, Madrid
Locations (1):
- UTRA and Clinica 4, at ULSSJOSÉ, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No
The security of personal and clinical data will be guaranteed, safeguarding the rights and freedoms of the data holder. The data collected will only be used for the purpose of this investigation, with access to them being exclusive to the researcher. The researcher will assume exclusive responsibility for processing and publishing the data, always seeking to preserve the identity of the participants. The data will only be kept for the time necessary to carry out the purpose of the investigation.